CLINICAL TRIAL: NCT00513526
Title: A Single-Arm, Open-Label Pilot Trial of the Safety and Immunogenicity of a Quadrivalent Human Papillomavirus Vaccine in HIV-1-Infected Men
Brief Title: Human Papillomavirus Vaccine Therapy in Treating Men With HIV-1 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-052; CDR0000559149 (Other: NCI); U01CA121947 (NIH)
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Results first posted 2011-07-26 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Infection; Precancerous Condition
Keywords: infection; low-grade squamous intraepithelial lesion; atypical squamous cells of undetermined significance
MeSH Terms: conditions — Infections; Precancerous Conditions; Squamous Intraepithelial Lesions; Atypical Squamous Cells of the Cervix | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gardasil (Experimental): Quadrivalent HPV Vaccine (types 6, 11, 16, 18) for intramuscular injection at study entry, week 8, week 24, and week 128.
  Interventions: Biological: Gardasil

INTERVENTIONS:
Biological: Gardasil — week 0, 8, 24, 128
  Other Names: quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine

SUMMARY:
RATIONALE: Vaccines made from human papillomavirus may help the body build an effective immune response to kill HIV cells.

PURPOSE: This phase II trial is studying the side effects and how well human papillomavirus vaccine therapy works in treating men with HIV-1 infection.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the safety and tolerability of quadrivalent human papillomavirus (HPV) (types 6, 11, 16, 18) recombinant vaccine in HIV-infected men.
* To assess the immunogenicity of the quadrivalent HPV vaccine for types 6, 11, 16 and 18 in subjects who are antibody-negative at baseline.

Secondary

* To evaluate the changes in plasma HIV-1 RNA and CD4+ count after the vaccination series.
* To describe the associations of CD4+ count, nadir CD4+ count, and age on antibody response.
* To evaluate the levels and persistence of HPV 6, 11, 16, and 18 antibody titers after the vaccination series among subjects according to serostatus at baseline.
* To evaluate the oral levels of serum IgA before and after the vaccination series.

Tertiary

* To evaluate prevalent and incident HPV infections in the anal canal.
* To evaluate cytological and histological abnormalities in the anal canal.
* To evaluate prevalent and incident HPV infections in the oral cavity.
* To compare oral and anal compartmental shedding of HPV before and after vaccination.

OUTLINE: This is a multicenter study.

Patients receive quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine intramuscularly on day 0 and weeks 8 and 24.

After completion of protocol therapy, patients are followed at 7, 12, and 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* HIV-1 infection, as documented by any licensed ELISA test kit and confirmed by western blot prior to study entry

  * HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test
* Anal human papilloma virus DNA PCR-negative for either type 16 and/or type 18 within 90 days prior to entry
* If receiving antiretroviral therapy:

  * Receipt of antiretroviral therapy for at least 6 months prior to entry
  * No change in antiretroviral therapy within 30 days prior to entry
  * CD4 cell count > 200 cells/mm³ within 90 days prior to study entry
  * HIV-1 RNA < 200 copies/mL within 90 days prior to entry
* If not receiving antiretroviral therapy:

  * CD4 cell count ≥ 350 cells/mm³ within 90 days prior to study entry
  * No plans to start antiretroviral therapy prior to week 28
* Normal anal cytological result, or atypical squamous cell of undetermined significance or low-grade squamous intraepithelial lesions (SIL) result within 90 days prior to entry

Exclusion criteria:

* Current or history of anal or perianal carcinoma
* Anal cytological result of high-grade SIL (HSIL), atypical squamous cells suggestive of HSIL, or suggestive of invasive carcinoma at screening or a history of these results
* Presence of high-grade anal intraepithelial neoplasm (HGAIN) (e.g., AIN 2 or 3, or perianal intraepithelial neoplasia grade 2 or 3), or invasive carcinoma at pre-entry, or history of HGAIN

  * Current or history of anal or peri-anal condyloma is allowed

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Karnofsky performance status 70-100%
* Absolute neutrophil count > 750 cells/mm³
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 100,000/mm³
* Creatinine clearance ≥ 60 mL/min
* AST and ALT ≤ 3 times ULN
* Total or conjugated (direct) bilirubin ≤ 2.5 times ULN

Exclusion criteria:

* Serious medical or psychiatric illness, active drug or alcohol use, or dependence that, in the opinion of the site Investigator, would interfere with adherence to study requirements
* Serious illness requiring systemic treatment and/or hospitalization within the past 45 days
* Allergy to yeast or any of the components of quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine
* Hemophilia

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* See Disease Characteristics

Exclusion criteria:

* Prior splenectomy
* Currently receiving anticoagulation therapy other than acetylsalicylic acid
* Use of any systemic antineoplastic or immunomodulatory treatment, systemic corticosteroids, investigational vaccines, interleukins, interferons, growth factors, or IVIG within 45 days prior to study entry

  * Routine standard of care, including hepatitis A or B, influenza, or pneumococcal and tetanus vaccines are not excluded
  * Hepatitis C co-infected patients are eligible provided no concurrent initiation of treatment for hepatitis C
* Prior receipt of quadrivalent HPV (types 6, 11, 16, 18) recombinant vaccine or other HPV vaccine

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2007-11; Primary Completion 2010-05 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J. Wilkin, MD, MPH, Study Chair — Weill Medical College of Cornell University; Joel Palefsky, MD, Principal Investigator — University of California, San Francisco
Locations (8):
- United States (8):
  - UCLA Clinical AIDS Research and Education (CARE) Center, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Denver Health Medical Center, Denver, Colorado
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Laser Surgery Care, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Benaroya Research Institute at Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Kang M, Umbleja T, Ellsworth G, Aberg J, Wilkin T. Effects of Sex, Existing Antibodies, and HIV-1-Related and Other Baseline Factors on Antibody Responses to Quadrivalent HPV Vaccine in Persons With HIV. J Acquir Immune Defic Syndr. 2022 Apr 1;89(4):414-422. doi: 10.1097/QAI.0000000000002891. PMID 34907980
- [Derived] Wilkin T, Lee JY, Lensing SY, Stier EA, Goldstone SE, Berry JM, Jay N, Aboulafia D, Cohn DL, Einstein MH, Saah A, Mitsuyasu RT, Palefsky JM. Safety and immunogenicity of the quadrivalent human papillomavirus vaccine in HIV-1-infected men. J Infect Dis. 2010 Oct 15;202(8):1246-53. doi: 10.1086/656320. PMID 20812850
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials/NCT00513526

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gardasil
Started | 109
Completed | 92
Not Completed | 17

BASELINE CHARACTERISTICS:
Arm/Group | Gardasil
Number analyzed (Participants) | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 109
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 109
Region of Enrollment [Number; unit: participants]
  United States | 109

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of ≥ Grade 3 Adverse Events Probably or Definitely Related to the Vaccine
Description: Occurrence of grade 3+ adverse events that are at least probably and definitely related to the vaccine
Time Frame: All study visits
Population: Intention to treat (i.e., received at least one dose of the vaccine)
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Gardasil: The single arm study is performed among HIV infected adult men satisfying the study eligibility criteria, including either PCR-negative for HPV 16 and/or HPV 18, or up to 20 subjects with PCR-positive for HPV 16 and HPV 18 each. Subjects are excluded if they have an anal cytology showing high-grade intraepithelial lesion(s) (HSIL), atypical squamous cells of undetermined significance (ASCUS) suggestive of HSIL or cytology suggestive of carcinoma. Subjects with a cytological result that is normal, ASCUS or low grade intraepithelial lesion(s) (LSIL) are eligible if subsequent anal biopsies obtained during high-resolution anoscopy at pre-entry show no evidence of HGAIN or squamous cell carcinoma. At study entry, subjects will give samples for HPV DNA PCR, and HPV type-specific serologies. Subjects will receive the HPV vaccine on Day 1, Week 8 and Week 24. Subsequently, subjects will be seen for study visits through 18 months after entry (12 months after vaccination). HPV DNA PCR, liquid based anal cytology, high resolution anoscopy with biopsy and HPV serologies (types 6, 11, 16 and 18) will be obtained during study follow-up
Arm/Group | Gardasil
Number analyzed (Participants) | 109
participants | 0 [NA to 0.0275] — Upper bound of confidence interval. No participant experienced grade 3 or greater events attributable to the vaccine

2. Primary Outcome: Detectable Human Papillomavirus (HPV) Antibody to Type 6 a Month After the Completion of HPV Vaccination Series (Week 28) Among Patients Seronegative for Type 6 at Baseline
Time Frame: Week 28
Population: Per protocol population for a given HPV type requires patients to be seronegative for that type at entry and to have no HPV DNA detected by PCR for that type at entry and screening. Also, patients must have received 3 doses of vaccine.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Gardasil: Number of participants seropositive for HPV-6 at week 28 among those who were seronegative at baseline.
Arm/Group | Gardasil
Number analyzed (Participants) | 60
proportion of participants | 0.98 [0.92 to NA] — Lower one-sided 95% confidence interval

3. Secondary Outcome: Longitudinal Changes in CD4+ Cell Count From Baseline
Description: CD4+ cell count at week 0 was subtracted from CD4+ cell counts at each of weeks 4, 12, and 28.
Time Frame: Week 0, 4, 12, 28
Population: Intention to treat population, includes all participants who received at least one dose of vaccine and had assessments at week 0 and the specified week.
Measure: Median (Inter-Quartile Range); unit: cells/uL
Groups:
- Gardasil: The enrolled subjects will receive Quadrivalent HPV (Types 6, 11, 16, 18) recombinant vaccine, 0.5 mL, intramuscularly in the deltoid region of the upper arm or the higher anterolateral area of the thigh on day 0, Week 8 and Week 24. A 4th dose will be given at week 128.
Arm/Group | Gardasil
Number analyzed (Participants) | 109
cells/uL
  Change from baseline at week 4 | 11 [-81 to 71]
  Change from baseline at week 12 | 9 [-56 to 70]
  Change from baseline at week 28 | 1 [-72 to 71]

4. Secondary Outcome: Longitudinal Changes in Plasma HIV-1 RNA From Baseline
Description: Plasma HIV-1 RNA at week 0 was subtracted from plasma HIV-1 RNA at each of weeks 4, 12, and 28.
Time Frame: Week 0, 4, 12, 28
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: copies/ml
Arm/Group | Gardasil
Number analyzed (Participants) | 103
copies/ml
  Baseline | 38 [24 to 94]
  Change at 4 weeks from the baseline: number analyzed (Participants) | 95
  Change at 4 weeks from the baseline | 0 [-1 to 0]
  Change at 12 weeks from the baseline: number analyzed (Participants) | 92
  Change at 12 weeks from the baseline | 0 [-1 to 0]
  Change at 28 weeks from the baseline: number analyzed (Participants) | 90
  Change at 28 weeks from the baseline | 0 [-1 to 12]

5. Secondary Outcome: HPV Antibody Titers to Type 6 at Baseline and Weeks 28 and 76 According to Baseline Seropositive Status
Description: HPV antibody titers to type 6 at baseline and weeks 28 and 76 according to baseline seropositive status will measured in Milli-Merck units per milliliters
Time Frame: weeks 0, 28, and 76
Population: Intent to treat population, includes all participants who received at least one dose of vaccine
Measure: Geometric Mean (95% Confidence Interval); unit: Milli-Merck units/mL
Arm/Group | Gardasil
Number analyzed (Participants) | 109
Milli-Merck units/mL
  Seropositive Group at Baseline | 76 [58 to 98]
  Seropositive Group at Week 28 | 933 [525 to 1657]
  Seropositive Group at Week 76 | 613 [393 to 959]
  Seronegative Group at Baseline | 5 [5 to 7]
  Seronegative Group at Week 28 | 336 [242 to 467]
  Seronegative Group at Week 76 | 146 [115 to 186]

6. Primary Outcome: Detectable Human Papillomavirus (HPV) Antibody to Type 11 a Month After the Completion of HPV Vaccination Series (Week 28) Among Patients Seronegative for Type 11 at Baseline
Time Frame: Week 28
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Gardasil
Number analyzed (Participants) | 68
proportion of participants | 0.99 [0.93 to NA] — Lower one-sided 95% confidence interval

7. Primary Outcome: Detectable Human Papillomavirus (HPV) Antibody to Type 16 a Month After the Completion of HPV Vaccination Series (Week 28) Among Patients Seronegative for Type 16 at Baseline
Time Frame: Week 28
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Gardasil
Number analyzed (Participants) | 62
proportion of participants | 1.00 [0.95 to NA] — Lower one-sided 95% confidence interval

8. Primary Outcome: Detectable Human Papillomavirus (HPV) Antibody to Type 18 a Month After the Completion of HPV Vaccination Series (Week 28) Among Patients Seronegative for Type 18 at Baseline
Time Frame: Week 28
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Gardasil
Number analyzed (Participants) | 77
proportion of participants | 0.95 [0.89 to NA] — Lower one-sided 95% confidence interval

9. Secondary Outcome: HPV Antibody Titers to Type 11 at Baseline and Weeks 28 and 76 According to Baseline Seropositive Status
Description: HPV antibody titers to type 11 at baseline and weeks 28 and 76 according to baseline seropositive status will measured in Milli-Merck units per milliliters
Time Frame: weeks 0, 28, and 76
Population: Intent to treat population, includes all participants who received at least one dose of vaccine
Measure: Geometric Mean (95% Confidence Interval); unit: Milli-Merck units/mL
Arm/Group | Gardasil
Number analyzed (Participants) | 109
Milli-Merck units/mL
  Seropositive Group at Baseline | 53 [42 to 66]
  Seropositive Group at Week 28 | 1536 [1089 to 2168]
  Seropositive Group at Week 76 | 797 [520 to 1221]
  Seronegative Group at Baseline | 5 [5 to 6]
  Seronegative Group at Week 28 | 503 [385 to 658]
  Seronegative Group at Week 76 | 196 [151 to 253]

10. Secondary Outcome: HPV Antibody Titers to Type 16 at Baseline and Weeks 28 and 76 According to Baseline Seropositive Status
Description: HPV antibody titers to type 16 at baseline and weeks 28 and 76 according to baseline seropositive status will measured in Milli-Merck units per milliliters
Time Frame: weeks 0, 28, and 76
Population: Intent to treat population, includes all participants who received at least one dose of vaccine
Measure: Geometric Mean (95% Confidence Interval); unit: Milli-Merck units/mL
Arm/Group | Gardasil
Number analyzed (Participants) | 109
Milli-Merck units/mL
  Seropositive Group at Baseline | 83 [59 to 117]
  Seropositive Group at Week 28 | 2005 [1215 to 3309]
  Seropositive Group at Week 76 | 1225 [779 to 1926]
  Seronegative Group at Baseline | 6 [5 to 6]
  Seronegative Group at Week 28 | 1001 [745 to 1346]
  Seronegative Group at Week 76 | 287 [202 to 408]

11. Secondary Outcome: HPV Antibody Titers to Type 18 at Baseline and Weeks 28 and 76 According to Baseline Seropositive Status
Description: HPV antibody titers to type 18 at baseline and weeks 28 and 76 according to baseline seropositive status will measured in Milli-Merck units per milliliters
Time Frame: weeks 0, 28, and 76
Population: Intent to treat population, includes all participants who received at least one dose of vaccine
Measure: Geometric Mean (95% Confidence Interval); unit: Milli-Merck units/mL
Arm/Group | Gardasil
Number analyzed (Participants) | 109
Milli-Merck units/mL
  Seropositive Group at Baseline | 53 [39 to 73]
  Seropositive Group at Week 28 | 765 [446 to 1313]
  Seropositive Group at Week 76 | 370 [202 to 679]
  Seronegative Group at Baseline | 5 [5 to 6]
  Seronegative Group at Week 28 | 181 [138 to 238]
  Seronegative Group at Week 76 | 38 [27 to 54]

12. Secondary Outcome: Evaluate Oral Levels of Serum IgA Before and After the Vaccination Series
Time Frame: Weeks 0, 28 and 76
Population: Samples for this outcome measure were not analyzed due to loss of funding for the central lab.
Arm/Group | Gardasil
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Gardasil
Serious Adverse Events (participants affected / at risk) | 5/109
Other Adverse Events (participants affected / at risk) | 56/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gardasil (N=109)
Hepatobiliary/Pancreas - Other (Specify, __) (Hepatobiliary disorders) | 1 (1)
Pain / Head/Headache (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Musculoskeletal/Soft Tissue - Other (Specifiy, __) (Musculoskeletal and connective tissue disorders) | 1 (2)
Infection with Normal ANC or Grade 1 or 2 Neutrophils/Bone (Osteomyelitis) (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gardasil (N=109)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Fatigue (Asthenia, Lethargy, Malaise) (General disorders) | 6 (6)
Infection - Other (Specify, __) (Infections and infestations) | 8 (9)
Infection with Normal ANC or Grade 1 or 2 Neutrophils / Upper Airway NOS (Infections and infestations) | 10 (11)
Infection with Unknown ANC / Upper Airway NOS (Infections and infestations) | 8 (9)
Injection Site Reaction / Extravasation Changes (Injury, poisoning and procedural complications) | 35 (62)
Pain - Other (Specifiy, __) (General disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No